CLINICAL TRIAL: NCT04483921
Title: Race Differences in 24-hour Energy Expenditure, Substrate Oxidation, and Appetite in Adolescent Girls
Brief Title: SubsTRate OxidatioN in Girls
Acronym: STRONG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Nutrition Obesity Research Center (Other)
Responsible Party: Principal Investigator, Eric Ravussin, Professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PBRC 2020-003
Record Dates: First submitted 2020-07-14; First posted 2020-07-23 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Overweight Adolescents
Keywords: Energy expenditure; Substrate oxidation; Appetite; Exercise; Energy intake
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Within-subjects crossover design. The order of conditions is counterbalanced within each subgroup of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Participants will complete a prescribed exercise bout.
  Interventions: Other: Acute exercise
- Sedentary (No Intervention): Participants will rest quietly in a seated position for the equivalent amount of time prescribed for the exercise condition.

INTERVENTIONS:
Other: Acute exercise — Participants will complete a morning exercise bout at 70% of their individual maximal aerobic capacity to burn 200 kilocalories above their basal metabolic rate.
  Arms: Exercise

SUMMARY:
This study will examine race differences in total energy expenditure and respiratory quotient (RQ) during and after exercise, compared to a sedentary control condition, in adolescent girls who are classified as overweight. In addition, subjective appetite and objective energy intake will be measured throughout the assessment periods.

DETAILED DESCRIPTION:
Aim 1: Measure 24-hour energy expenditure and its components (resting, activity, and sleep energy expenditure) and compare differences between African-American and White girls.

Hypothesis: Total, resting, and sleep energy expenditure will be lower in African-American relative to White girls. Activity energy expenditure will be equivalent per the study design.

Aim 2: Measure and compare substrate oxidation and associations with appetite (i.e., hunger, desire to eat) and energy intake between African-American and White girls.

Hypothesis: African-American girls will have a higher RQ at rest, during exercise, and following exercise, and RQ will be positively associated with subjective appetite ratings and energy intake.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 13-17 years, inclusive
* Achieved menarche based on parent- and/or self-report
* Overweight based on BMI percentile for age and sex (≥ 85th and < 95th)
* Self-identification as non-Hispanic White or African-American
* Willing to maintain current physical activity, sleep schedule, and dietary habits during the study
* Willing to comply with study procedures

Exclusion Criteria:

* Contraindications to exercise testing as defined by the American College of Sports Medicine (i.e., medical history of cardiovascular, pulmonary, or physical conditions that affect the ability to exercise)
* Food allergies
* Dietary restrictions
* Unwilling to consume study foods
* History of polycystic ovary syndrome (PCOS)
* Current amenorrhea or other menstrual cycle irregularities
* Pregnant or currently breastfeeding
* Current anemia
* Use of medications affecting metabolism or sleep
* Inability to properly or safely complete the study procedures per the investigators' discretion

Ages: 13 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2023-09-02 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Exercise Day Energy expenditure | 24 hours on Exercise Day
  Total energy expenditure and its components (sleeping, wake [non-exercise], activity) as measured by the metabolic chamber
Sedentary Day Energy expenditure | 24 hours on Sedentary Day
  Total energy expenditure and its components (sleeping, wake [non-exercise], activity) as measured by the metabolic chamber
Exercise Day Substrate oxidation | 24 hours on Exercise Day
  Non-protein respiratory quotient (i.e., carbohydrate and fat utilization) as measured by the metabolic chamber
Sedentary Day Substrate oxidation | 24 hours on Sedentary Day
  Non-protein respiratory quotient (i.e., carbohydrate and fat utilization) as measured by the metabolic chamber

SECONDARY OUTCOMES:
Exercise Day Appetite | 24 hours on Exercise Day
  Overall subjective appetite and its components (hunger, fullness, desire to eat, prospective food consumption, satisfaction, food wanting) assessed by visual analog scales (0-100 mm) during the metabolic chamber assessments
Sedentary Day Appetite | 24 hours on Sedentary Day
  Overall subjective appetite and its components (hunger, fullness, desire to eat, prospective food consumption, satisfaction, food wanting) assessed by visual analog scales (0-100 mm) during the metabolic chamber assessments
Exercise Day Energy Intake | 24 hours on Exercise Day
  Objectively measured food intake during the metabolic chamber assessments will be converted to energy intake in kilocalories
Sedentary Day Energy Intake | 24 hours on Sedentary Day
  Objectively measured food intake during the metabolic chamber assessments will be converted to energy intake in kilocalories

OTHER OUTCOMES:
Dual-energy x-ray absorptiometry (DXA) | Baseline screening visit
  Total body composition (fat, muscle, bone tissue) measured by Hologic Discovery DXA
Body shape | Baseline screening visit
  3D optical imaging assessment of body shape by Fit3D scanner
Cardiorespiratory fitness | Baseline screening visit
  Maximal aerobic capacity assessed by graded cycle ergometer test to volitional fatigue
Resting metabolic rate | Baseline screening visit
  Measured over a 30-minute period by ventilated hood and metabolic cart
Implicit activity preferences | Baseline screening visit
  Relative preference for physical versus sedentary activities as assessed by a forced-choice behavioral task
Habitual physical activity | 7 days leading up to Exercise Day and Sedentary Day
  Accelerometry measures of usual physical activity before each experimental visit
Habitual sedentary time | 7 days leading up to Exercise Day and Sedentary Day
  Accelerometry measures of usual sedentary time before each experimental visit
Habitual food intake | 3 days leading up to Exercise Day and Sedentary Day
  Food intake diary/dietary record to assist participants in maintaining consistent diet before each experimental visit

CONTACTS AND LOCATIONS:
Overall Officials: Eric Ravussin, PhD, Principal Investigator — Professor
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
De-identified IPD will be housed indefinitely on secure digital servers as part of the Pennington Biomedical Clinical Database. De-identified IPD may be made available to other researchers upon reasonable request to the Principal Investigator, following Pennington Biomedical's standard procedures for data use agreements and secure data transfers.